CLINICAL TRIAL: NCT01652040
Title: Effects of Evoked Resistance Training and Testosterone After Spinal Cord Injury
Brief Title: Resistance Training and Testosterone After Spinal Cord Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: B7867-W
Record Dates: First submitted 2012-07-13; First posted 2012-07-27 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Rehabilitation; Electrical Stimulation; Testosterone; Body Composition; Lipid and Glucose profile; Ectopic Adiposity
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- RT+Tp (Experimental): Resistance training using electrical stimulation and ankle weights and Testosterone patches
  Interventions: Device: Resistance Training and Testosterone Patches
- Tp (Experimental): Applying Testosterone patches
  Interventions: Drug: Testosterone Patches

INTERVENTIONS:
Device: Resistance Training and Testosterone Patches — We are going to activate the knee extensor muscle group to lift ankle weights over 16 weeks and we are going to provide Tp to improve anabolic profile.
  Arms: RT+Tp
Drug: Testosterone Patches — The investigators will provide Tp patches for 16 weeks for patients with Spinal Cord Injury.
  Arms: Tp

SUMMARY:
The goal of this proposal is to investigate the efficacy of a complimentary approach of evoked resistance training and testosterone replacement therapy on the changes in body composition and metabolic profile after SCI. The proposed method could become a recommended and simple intervention especially for individuals with limited access and poor tolerance to exercise. The rationale is based on the evidence that individuals with SCI experience decline in anabolic hormones which may be responsible for the deterioration in body composition and metabolic profiles and leads to increase obesity, type 2 diabetes mellitus, dyslipidemia and subsequently cardiovascular disease. The designed study will provide explanation to the adaptations in the energy source of the muscle cells in response to training.

DETAILED DESCRIPTION:
Individuals with spinal cord injury (SCI) are at a lifelong risk of increasing obesity and several chronic metabolic disorders such as glucose intolerance, insulin resistance and dyslipidemia secondary to deterioration in body composition. Within few weeks of injury, there are significant decrease in whole body fat-free mass (FFM), particularly lower extremity skeletal muscle mass and subsequent increase in fat mass (FM). Resistance training (RT) is an important type of exercise that has been shown to induce positive physiological adaptations such as increasing lean mass and reducing metabolic disorders in other clinical populations.

In a pilot work, the investigators provided evidence that evoked RT using surface neuromuscular electrical stimulation (NMES) for knee extensor muscle group resulted in significant increase skeletal muscle cross-sectional area (CSA), reduction in % leg FM and a trend towards decrease in visceral adipose tissue (VAT) CSA. The favorable adaptations in body composition were associated with decrease in plasma insulin area under the curve and plasma triglycerides. The investigators attributed the adaptations in body composition and metabolic profile to an associated increase in plasma insulin-like growth factor (IGF-1). The investigators concluded that twelve weeks of evoked RT targeted towards evoking skeletal muscle hypertrophy could result in significant body composition and metabolic adaptations in individuals with SCI.

It is unclear if a longer RT program greater than 12 weeks would provide additional benefits to Veterans with SCI. It is also unknown whether enhancing the decline anabolic homeostasis by providing testosterone (T) replacement therapy (TRT) would reverse body composition and metabolic profile changes in Veterans with SCI. The major research goal of this proposal is to investigate the effects of 16 weeks of evoked RT+TRT vs. TRT on body composition (muscle CSA, VAT, %FM) and the metabolic profiles (glucose and lipid metabolism) in individuals with motor complete SCI. To address this goal, surface NMES accompanied with ankle weights will be conducted twice weekly to exercise the knee extensor skeletal muscle groups from sitting position. After 4 weeks of delayed entry approach, participants (n =24) will be randomly assigned into RT+TRT (n =12) or TRT (n =12) groups. The TRT will be provided via transdermal T patches that will be alternated on both shoulders over the course of the study. The investigators also propose to study the effects of detraining on body composition and metabolic profiles.

The research plan includes three specific aims

Specific aim 1 will demonstrate the effects of NMES RT and/or Testosterone patches (Tp) on the CSA of thighs and legs skeletal muscle groups, percentage FFM, and the CSA of VAT, intramuscular fat and percentage FM after 16 weeks of training+Tp and 16 weeks of detraining.

Specific aim 2 will determine the changes in metabolic milieu (resting energy expenditure, glucose homeostasis, lipid profile, free fatty acids, serum total and free testosterone and IGF-1), and cytokines (c-reactive protein, tumor necrosis factor alpha and IL-6 as inflammatory biomarkers) after 16 weeks of training+Tp and detraining.

Specific aim 3 will determine if 16 weeks of evoked RT and Tp will increase GLUT-4 concentration, muscle IGF-1 and peroxisome-proliferator-activated receptor-gamma co-activator 1 (PGC-1) expressions, altered fiber type distribution and enhance the mitochondrial enzymatic activities (electron transport chain) compared to Tp only.

ELIGIBILITY:
Inclusion Criteria:

* Male with Spinal Cord Injury
* Between 18-50 years old
* BMI < 30 Kg/m2
* Traumatic motor complete C5-L2 level of injury
* American Spinal Injury Classification (A and B; i.e. motor deficit below the level of injury)

Exclusion Criteria:

* Cardiovascular disease
* Uncontrolled type II DM and those on insulin
* Pressures sores stage 2 or greater
* Supra-physiological T level
* Hematocrit above 50%
* Urinary tract infection or symptoms

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Gorgey, PhD PT, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gorgey AS, Khalil RE, Gill R, O'Brien LC, Lavis T, Castillo T, Cifu DX, Savas J, Khan R, Cardozo C, Lesnefsky EJ, Gater DR, Adler RA. Effects of Testosterone and Evoked Resistance Exercise after Spinal Cord Injury (TEREX-SCI): study protocol for a randomised controlled trial. BMJ Open. 2017 Apr 4;7(4):e014125. doi: 10.1136/bmjopen-2016-014125. PMID 28377392
- [Background] Gorgey AS, Moore PD, Wade RC, Gill RS, Lavis T, Adler RA. Disruption in bone marrow fat may attenuate testosterone action on muscle size after spinal cord injury: a case report. Eur J Phys Rehabil Med. 2017 Aug;53(4):625-629. doi: 10.23736/S1973-9087.17.04452-5. Epub 2017 Mar 13. PMID 28290190
- [Background] Wade RC, Gorgey AS. Anthropometric prediction of skeletal muscle cross-sectional area in persons with spinal cord injury. J Appl Physiol (1985). 2017 May 1;122(5):1255-1261. doi: 10.1152/japplphysiol.01042.2016. Epub 2017 Mar 2. PMID 28255089
- [Background] O'Brien LC, Wade RC, Segal L, Chen Q, Savas J, Lesnefsky EJ, Gorgey AS. Mitochondrial mass and activity as a function of body composition in individuals with spinal cord injury. Physiol Rep. 2017 Feb;5(3):e13080. doi: 10.14814/phy2.13080. PMID 28193782
- [Background] Moore PD, Gorgey AS, Wade RC, Khalil RE, Lavis TD, Khan R, Adler RA. Neuromuscular electrical stimulation and testosterone did not influence heterotopic ossification size after spinal cord injury: A case series. World J Clin Cases. 2016 Jul 16;4(7):172-6. doi: 10.12998/wjcc.v4.i7.172. PMID 27458592
- [Background] Gorgey AS, Caudill C, Khalil RE. Effects of once weekly NMES training on knee extensors fatigue and body composition in a person with spinal cord injury. J Spinal Cord Med. 2016;39(1):99-102. doi: 10.1179/2045772314Y.0000000293. Epub 2015 Jan 23. PMID 25615403
- [Background] Gorgey AS, Mather KJ, Cupp HR, Gater DR. Effects of resistance training on adiposity and metabolism after spinal cord injury. Med Sci Sports Exerc. 2012 Jan;44(1):165-74. doi: 10.1249/MSS.0b013e31822672aa. PMID 21659900
- [Background] Gorgey AS, Shepherd C. Skeletal muscle hypertrophy and decreased intramuscular fat after unilateral resistance training in spinal cord injury: case report. J Spinal Cord Med. 2010;33(1):90-5. doi: 10.1080/10790268.2010.11689681. PMID 20397451
- [Background] Khalil RE, Gorgey AS, Janisko M, Dolbow DR, Moore JR, Gater DR. The role of nutrition in health status after spinal cord injury. Aging Dis. 2013 Feb;4(1):14-22. Epub 2012 Nov 30. PMID 23423356
- [Background] Gorgey AS, Dolbow DR, Cifu DX, Gater DR. Neuromuscular electrical stimulation attenuates thigh skeletal muscles atrophy but not trunk muscles after spinal cord injury. J Electromyogr Kinesiol. 2013 Aug;23(4):977-84. doi: 10.1016/j.jelekin.2013.04.007. Epub 2013 May 15. PMID 23683374
- [Background] Nightingale TE, Moore P, Harman J, Khalil R, Gill RS, Castillo T, Adler RA, Gorgey AS. Body composition changes with testosterone replacement therapy following spinal cord injury and aging: A mini review. J Spinal Cord Med. 2018 Nov;41(6):624-636. doi: 10.1080/10790268.2017.1357917. Epub 2017 Aug 3. PMID 28770686
- [Background] Gorgey AS, Lester RM, Wade RC, Khalil RE, Khan RK, Anderson ML, Castillo T. A feasibility pilot using telehealth videoconference monitoring of home-based NMES resistance training in persons with spinal cord injury. Spinal Cord Ser Cases. 2017 Jun 29;3:17039. doi: 10.1038/scsandc.2017.39. eCollection 2017. PMID 29021917
- [Background] Nightingale TE, Gorgey AS. Predicting Basal Metabolic Rate in Men with Motor Complete Spinal Cord Injury. Med Sci Sports Exerc. 2018 Jun;50(6):1305-1312. doi: 10.1249/MSS.0000000000001548. PMID 29315167
- [Background] Abilmona SM, Gorgey AS. Associations of the trunk skeletal musculature and dietary intake to biomarkers of cardiometabolic health after spinal cord injury. Clin Physiol Funct Imaging. 2018 Feb 6. doi: 10.1111/cpf.12505. Online ahead of print. PMID 29405604
- [Background] Rankin KC, O'Brien LC, Gorgey AS. Quantification of trunk and android lean mass using dual energy x-ray absorptiometry compared to magnetic resonance imaging after spinal cord injury. J Spinal Cord Med. 2019 Jul;42(4):508-516. doi: 10.1080/10790268.2018.1438879. Epub 2018 Feb 20. PMID 29461936
- [Background] McCauley LS, Sumrell RM, Gorgey AS. Anthropometric Prediction of Visceral Adipose Tissue in Persons With Motor Complete Spinal Cord Injury. PM R. 2018 Aug;10(8):817-825.e2. doi: 10.1016/j.pmrj.2018.02.007. Epub 2018 Feb 21. PMID 29474998
- [Background] Gorgey AS, Cirnigliaro CM, Bauman WA, Adler RA. Estimates of the precision of regional and whole body composition by dual-energy x-ray absorptiometry in persons with chronic spinal cord injury. Spinal Cord. 2018 Oct;56(10):987-995. doi: 10.1038/s41393-018-0079-x. Epub 2018 Mar 6. PMID 29511310
- [Background] O'Brien LC, Graham ZA, Chen Q, Lesnefsky EJ, Cardozo C, Gorgey AS. Plasma adiponectin levels are correlated with body composition, metabolic profiles, and mitochondrial markers in individuals with chronic spinal cord injury. Spinal Cord. 2018 Sep;56(9):863-872. doi: 10.1038/s41393-018-0089-8. Epub 2018 Mar 20. PMID 29559683
- [Result] O'Brien LC, Chen Q, Savas J, Lesnefsky EJ, Gorgey AS. Skeletal muscle mitochondrial mass is linked to lipid and metabolic profile in individuals with spinal cord injury. Eur J Appl Physiol. 2017 Nov;117(11):2137-2147. doi: 10.1007/s00421-017-3687-9. Epub 2017 Sep 1. PMID 28864949
- [Result] Rankin KC, O'Brien LC, Segal L, Khan MR, Gorgey AS. Liver Adiposity and Metabolic Profile in Individuals with Chronic Spinal Cord Injury. Biomed Res Int. 2017;2017:1364818. doi: 10.1155/2017/1364818. Epub 2017 Aug 30. PMID 28948164
- [Derived] Gorgey AS, Khalil RE, Gill R, Khan R, Adler RA. Effects of dose de-escalation following testosterone treatment and evoked resistance exercise on body composition, metabolic profile, and neuromuscular parameters in persons with spinal cord injury. Physiol Rep. 2021 Nov;9(21):e15089. doi: 10.14814/phy2.15089. PMID 34713983
- [Derived] Holman ME, Chang G, Ghatas MP, Saha PK, Zhang X, Khan MR, Sima AP, Adler RA, Gorgey AS. Bone and non-contractile soft tissue changes following open kinetic chain resistance training and testosterone treatment in spinal cord injury: an exploratory study. Osteoporos Int. 2021 Jul;32(7):1321-1332. doi: 10.1007/s00198-020-05778-2. Epub 2021 Jan 14. PMID 33443609
- [Derived] Gorgey AS, Graham ZA, Chen Q, Rivers J, Adler RA, Lesnefsky EJ, Cardozo CP. Sixteen weeks of testosterone with or without evoked resistance training on protein expression, fiber hypertrophy and mitochondrial health after spinal cord injury. J Appl Physiol (1985). 2020 Jun 1;128(6):1487-1496. doi: 10.1152/japplphysiol.00865.2019. Epub 2020 Apr 30. PMID 32352341
- [Derived] Holman ME, Gorgey AS. Testosterone and Resistance Training Improve Muscle Quality in Spinal Cord Injury. Med Sci Sports Exerc. 2019 Aug;51(8):1591-1598. doi: 10.1249/MSS.0000000000001975. PMID 30845047
- [Derived] Gorgey AS, Khalil RE, Gill R, Gater DR, Lavis TD, Cardozo CP, Adler RA. Low-Dose Testosterone and Evoked Resistance Exercise after Spinal Cord Injury on Cardio-Metabolic Risk Factors: An Open-Label Randomized Clinical Trial. J Neurotrauma. 2019 Sep 15;36(18):2631-2645. doi: 10.1089/neu.2018.6136. Epub 2019 Mar 28. PMID 30794084

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Replacement Patches (Tp): Applying Testosterone patches
  Testosterone Patches: The investigators will provide Tp patches for 16 weeks for patients with Spinal Cord Injury.
Period: Overall Study
Arm/Group | RT+Tp | Testosterone Replacement Patches (Tp)
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Persons with motor complete AIS A or B and level of injury C5 and with age under 50 years old.
Groups:
- Total: Total of all reporting groups
Arm/Group | RT+Tp | Testosterone Replacement Patches (Tp) | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12) | 35 (8) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: Changes in body composition fat mass
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of fat mass
Groups:
- Testosteroe Replacement Patches (Tp): Applying Testosterone patches
  Testosterone Patches: The investigators will provide Tp patches for 16 weeks for patients with Spinal Cord Injury.
Arm/Group | RT+Tp | Testosteroe Replacement Patches (Tp)
Number analyzed (Participants) | 11 | 11
percentage of fat mass
  Baseline | 31.84 (10.7) | 33.4 (9)
  Post-Intervention (After 16 weeks) | 30.75 (10.3) | 32.12 (9)

2. Secondary Outcome: Metabolic Profile
Description: Basal Metabolic Rate
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | RT+Tp | Testosterone Replacement Patches (Tp)
Number analyzed (Participants) | 11 | 11
kcal/day
  Baseline | 1525 (261) | 1491 (177)
  Post-Intervention (After 16 weeks) | 1665 (243) | 1502 (327)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse Events were monitored for skin irritation from using testosterone patches
Arm/Group | RT+Tp | Testosterone Replacement Patches (Tp)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT01652040/Prot_SAP_000.pdf